CLINICAL TRIAL: NCT03080558
Title: Estimation of Vascularization After Treatment of Deep Rectovaginal Endometriosis Node by Rectal Shaving, Using Indocyanine Green Injection. Feasibility Study
Brief Title: Estimation of Vascularization After Treatment of Deep Rectovaginal Endometriosis Node by Rectal Shaving
Acronym: INDIE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire SERB (Unknown); Association GEGO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-305; 2016-002773-35 (Other: 2016-002773-35)
Record Dates: First submitted 2017-03-06; First posted 2017-03-15 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Deep Endometriosis; Recto Vaginal Node
Keywords: Indocyanine green fluorescence; Rectal vascularisation; Vaginal vascularisation; Laparoscopic surgery; Rectal shaving; Recto vaginal node; Deep Endometriosis
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endometriosis recto vaginal node (Experimental)
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Use of Indocyanine Green during Rectal shaving by laparoscopy.

SUMMARY:
Indocyanine green is a dye, using in surgery to bring out the intraoperative evaluation of tissue perfusion.

After intravenous injection of indocyanine green, using a near infrared light, the vascularisation becomes fluorescent.

In endometriosis disease, the treatment of recto vaginal node can be complicated by rectovaginal fistula.

An abnormal vascularisation related to the surgery would be a risk factor of post operative fistulas.

The aim of this study is to evaluate the rectal and vaginal vascularisation during the treatment of a recto vaginal endometriosis nodule with rectal shaving, using indocyanine green fluorescence.

DETAILED DESCRIPTION:
Investigators are going to inject, at the end of a rectal shaving, a bolus of 0,2mg/kg of indocyanine green after dilution (2,5mg/ml). With de SPIES system (KARL STORZ GmbH & Co. KG, Tuttlingen, Germany), the vascularisation would be imediately fluorescent. Investigators are going to estimate the vascularization of the rectal serosa and mucosa where the nodule was located.

If a vaginal resection has been performed, investigators are going to estimate the vascularization of the vaginal scar.

To estimate de vascularization, investigators are going tu use a scale with a score between 0 and 4.

After the surgery, the post-operative follow-up with be the same as usual after a Rectal Shaving.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 year
* Patients with endometriosis recto vaginal node
* Patients with operative indications of rectal shaving, with or without vaginal resection
* Patients who have accepted to participate

Exclusion Criteria:

* minors patients
* Patients under guardianship or wardship
* Patients who refused the participation
* Iodine allergy
* Pregnant woman
* Patients during lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-06 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Per-operative evaluation of the rectum | at day 1
  Per-operative evaluation of the rectum after Shaving, using indocyanine green fluorescence, by transperitoneal and intra-rectal approach, and vaginal suture if there is an associated vaginal resection. A fluorescence score between 0 and 4 will be used, based on a Likert scale

SECONDARY OUTCOMES:
Side effects after indocyanine green injection | at day 1
Post operative complications | at day 1
  infections, abdominal abscess, abdominal hematoma, post operative fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BOURDEL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Bourdel N, Jaillet L, Bar-Shavit Y, Comptour A, Pereira B, Canis M, Chauvet P. Indocyanine green in deep infiltrating endometriosis: a preliminary feasibility study to examine vascularization after rectal shaving. Fertil Steril. 2020 Aug;114(2):367-373. doi: 10.1016/j.fertnstert.2020.03.042. Epub 2020 Jul 7. PMID 32646588
- [Derived] Bar-Shavit Y, Jaillet L, Chauvet P, Canis M, Bourdel N. Use of indocyanine green in endometriosis surgery. Fertil Steril. 2018 Jun;109(6):1136-1137. doi: 10.1016/j.fertnstert.2018.02.113. Epub 2018 Jun 6. PMID 29885885